CLINICAL TRIAL: NCT04471753
Title: Target Behaviours to Identify Minimally Conscious State Patients by Using Coma Recovery Scale-Revised
Brief Title: Target Behaviours to Identify Minimally Conscious State Patients
Status: Completed | Type: Observational
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Jing Wang, Principal Investigator, Hangzhou Normal University
Other Study IDs: 2020N39286
Record Dates: First submitted 2020-07-12; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Disorder of Consciousness; Minimally Conscious State
Keywords: disorders of consciousness; Coma Recovery Scale-revision; minimally conscious state
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with disorders of consciousness: Patients with medical diagnosis of prolonged disorders of consciousness (≥28 days) were included in neurosurgery, neurology, and neurorehabilitation units.
  Interventions: Behavioral: Coma Recovery Scale-Revised

INTERVENTIONS:
Behavioral: Coma Recovery Scale-Revised — Data were collected according to the Coma Recovery Scale-Revised operation guideline, the sum of the highest score on the evaluated subscales was taken as the final score, and the final diagnosis of patients was obtained (the highest score of each subscale was recorded). All participants were diagnosed by using CRS-R five times at least within 7 days. According to the results of the Coma Recovery Scale-Revised assessment, minimally conscious state and unresponsive wakefulness syndrome were distinguished.

SUMMARY:
To analyse the frequency of the consciousness behaviour response for patients with minimally conscious state of Coma Recovery Scale-Revised items, as well as the necessary items for obtaining higher accuracy. In addition, providing target behaviours for Coma Recovery Scale-Revised assessment of minimally conscious state diagnosis and evidence for the simplification of Coma Recovery Scale-Revised in the future.

DETAILED DESCRIPTION:
Data were collected according to the Coma Recovery Scale-Revised operation guideline, the sum of the highest score on the evaluated subscales was taken as the final score, and the final diagnosis of patients was obtained (the highest score of each subscale was recorded). All participants were diagnosed by using Coma Recovery Scale-Revised five times at least within 7 days. According to the results of the Coma Recovery Scale-Revised assessment, minimally conscious state and unresponsive wakefulness syndrome patients were distinguished.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medical diagnosis of prolonged disorders of consciuosness (≥28 days) were included in neurosurgery, neurology, and neurorehabilitation units.

Exclusion Criteria:

* Patients who used neuromuscular blockers or sedatives within 72 hours of enrolment were excluded.

Ages: 18 Years to 84 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients were assessed by the Coma Recovery Scale-Revised for several times with seven days.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised | Within 7 days
  The Coma Recovery Scale-Revised has 23 items, which evaluate the patients' auditory, visual, motor, oromotor/verbal, communication, and arousal functions. For each subscale, the lower score reflects reflexivity related to the brain stem, while the higher score reflects non-reflexivity related to higher cortical functions.

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Di, Pro., Study Chair — Hangzhou Normal University
Locations (1):
- International Vegetative State and Consciousness Science Institute, Hangzhou Normal University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Wannez S, Heine L, Thonnard M, Gosseries O, Laureys S; Coma Science Group collaborators. The repetition of behavioral assessments in diagnosis of disorders of consciousness. Ann Neurol. 2017 Jun;81(6):883-889. doi: 10.1002/ana.24962. PMID 28543735
- [Result] American Congress of Rehabilitation Medicine, Brain Injury-Interdisciplinary Special Interest Group, Disorders of Consciousness Task Force; Seel RT, Sherer M, Whyte J, Katz DI, Giacino JT, Rosenbaum AM, Hammond FM, Kalmar K, Pape TL, Zafonte R, Biester RC, Kaelin D, Kean J, Zasler N. Assessment scales for disorders of consciousness: evidence-based recommendations for clinical practice and research. Arch Phys Med Rehabil. 2010 Dec;91(12):1795-813. doi: 10.1016/j.apmr.2010.07.218. PMID 21112421